CLINICAL TRIAL: NCT03991702
Title: Hand Grip Strength and Medical Research Council Scale as Predictors of Weaning Failure and Duration of Mechanical Ventilation.
Brief Title: Hand Grip Strength and Medical Research Council Scale as Predictors of Weaning Failure
Status: Completed | Type: Observational
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Other Study IDs: 49900015.0.0000.5327
Record Dates: First submitted 2019-05-29; First posted 2019-06-19 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Muscle Weakness Condition; Mechanical Ventilation Complication; Weaning Failure
MeSH Terms: interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: diagnostic test — The overall motor function of the patient will be assessed using the Medical Research Council (MRC) scale and Palmar dynamometer strength

SUMMARY:
The handgrip strength (HGS) will be measured with a digital dynamometer. Three measurements will be taken, whose average of the three measurements will be collected.

Muscle weakness will be diagnosed based on previously published ICU acquired weakness (ICU-AW) scores (for males <11 kg and females <7 kg).

The overall motor function of the patient will be assessed using the Medical Research Council (MRC) scale. The maximum score of the scale is 60 points, adding the degree of muscle strength of all muscle groups tested. If the patient is unable to have one of the limbs tested, it is assumed that the limb would have the same force as the contralateral limb.

A score of 48 points or less is indicative of muscle weakness. Individuals who scored between 48 and 37 points on the MRC scale are considered to have significant weaknesses; those with 36 points or less are classified as severely weak.

The HGS and the MRC scale will be compared as predictors of weaning duration of mechanical ventilation

DETAILED DESCRIPTION:
The handgrip strength will be measured with a digital dynamometer. The patient's dominant hand will be tested, with the patient as seated as possible, with the elbow as close as to 90º. Three measurements will be taken, respecting a minute interval between them, whose average of the three measurements will be collected.

Muscle weakness will be diagnosed based on previously published weakness scores (for males <11 kg (kilograms) and females <7 kg) 25. The strength value will be normalized as a relative value in percent, calculated according to Bohannon et al. based on values of healthy individuals, considering gender and age. It will also be normalized according to height, due to the known impact of this anthropometric feature on palmar strength.

The overall motor function of the patient will be assessed using the Medical Research Council (MRC) 24 scale. The evaluation will consist of the bilateral analysis of six specific movements (shoulder abduction, elbow flexion, wrist flexion, hip flexion, knee extension, ankle dorsiflexion) through manual muscle testing, scoring from zero to five points 2 = movement without the action of gravity, 3 = movement against the action of gravity, 4 = a slight manual resistance wins, 5 = a great manual resistance wins ). The maximum score of the scale is 60 points, adding the degree of muscle strength of all muscle groups tested. If the patient is unable to have one of the limbs tested (for example: amputation) it is assumed that the limb would have the same force as the contralateral limb.

In order to standardize the position during the application of the scale and to minimize bias, the position will be adopted in the supine position, with the bed between 45º to 60º and symmetrical posture. First the patient will be asked to move freely. According to the result, manual resistance is imposed or the action of gravity is eliminated.

The indicative weakness score is 48 points or less. Individuals who score between 48 and 37 points on the MRC scale are considered to have significant weaknesses; those with 36 points or less are classified as severely weak.

The handgrip strength and the MRC scale will be compared as predictors of weaning duration of mechanical ventilation

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* being on invasive mechanical ventilation for more than 48 hours
* fulfill the pre-defined criteria for performing the spontaneous breathing test

Exclusion Criteria:

- patients unable to perform the hand grip strength test and the MRC scale (any rheumatologic conditions, neuromuscular, amputation, cachexia, neuropsychiatric symptoms: such as confusion and delirium)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients on invasive mechanical ventilation for more than 48 hours and ready to perform the spontaneous breathing test.
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
mechanical ventilation weaning time | 30 days
  to evaluate the hand grip strength as a predictor of spontaneous breathing test failure and the duration of mechanical ventilation weaning.
Duration of mechanical ventilation | 30 days
  to evaluate the Medical Research Council scale as a predictor of spontaneous breathing test failure and the duration of mechanical ventilation. The MRC score is obtained by evaluating 12 muscle groups in the upper extremities (wrist extensors, elbow flexors and abductors of the shoulder) and lower extremities (dorsal ankle flexors, knee extensors, and hip flexors). For each muscle group will be assigned a score between 0 (complete paralysis) and 5 (normal force), and the total score can vary between 0 up to 60 points.

SECONDARY OUTCOMES:
HGS cut-off points indicative of ICU acquired Weakness | 30 days
  to define HGS cut-off points indicative of ICU acquired weakness for men and women

CONTACTS AND LOCATIONS:
Overall Officials: Gilberto Friedman, Prof, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No